CLINICAL TRIAL: NCT04900935
Title: Patient-centered, Optimal Integration of Survivorship and Palliative Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura Petrillo, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-722; K08CA263549 (NIH)
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Stage IV Non-small Cell Lung Cancer; Targeted Therapy; Nonsmall Cell Lung Cancer; Carcinoma, Non-Small-Cell Lung; ALK-positive Non-small Cell Lung Cancer; EGFR Positive Non-small Cell Lung Cancer; Palliative Care; Survivorship
Keywords: Stage IV Non-small Cell Lung Cancer; Targeted Therapy; Nonsmall Cell Lung Cancer; Carcinoma, Non-Small-Cell Lung; ALK-positive Non-small Cell Lung Cancer; EGFR Positive Non-small Cell Lung Cancer; ROS1 Positive Non-Small Cell Lung Cancer; Palliative care; survivorship; RET Fusion positive Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: There will be two phases of this research study: 1) an open pilot of 10 patients to refine the intervention and study protocol, in which all patients receive the POISE intervention; followed by 2) a randomized controlled trial in which patients are randomized to receive either the POISE intervention or usual care.
Who Masked: Outcomes Assessor
Masking Description: Masking of participants and care providers is not possible in this clinical intervention. However, we will mask the outcomes assessor to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- POISE (Experimental): The intervention will be a structured palliative care intervention in which patients will meet with a palliative care clinician who has been trained on a manual with specific topics to be covered in each of the four visits:
  * Three surveys: baseline, 12-week, and 20-week post-enrollment
  * Four 60-minute visits with a trained palliative care clinician
  * Semi-structured exit interview
  * Chart review
  Interventions: Behavioral: POISE
- Usual care (No Intervention): Patients randomized to usual care will receive usual oncology care. They may access standard palliative care as clinically indicated.

INTERVENTIONS:
Behavioral: POISE — POISE (Patient-centered, Optimal Integration of Survivorship and palliative carE) is a brief, population-specific intervention that consists of four sessions with palliative care specialists who have been additionally trained to evaluate and address the specific psychosocial issues and health-promoting behaviors of patients with long, uncertain cancer trajectories.
  Other Names: palliative care intervention
  Arms: POISE

SUMMARY:
The goal of this study is to develop and test the feasibility of a supportive care model (POISE) for patients with metastatic Non-small Cell Lung Cancer (NSCLC). The main questions are

* is POISE feasible to deliver and acceptable to patients
* what is the effect of POISE on the distress patients feel related to their uncertain future, their confidence in their ability to manage cancer, and their understanding about what to expect Participants in the randomized controlled trial will receive either the new supportive care model, POISE, which consists of four visits with a trained palliative care clinician, or care as usual, and will be asked to complete three surveys.

DETAILED DESCRIPTION:
This research study involves an intervention consisting of four sessions with palliative care specialists who have been additionally trained to evaluate and address the specific psychosocial issues and health-promoting behaviors of patients with NSCLC.

The research study procedures include:

* Four 60-minute visits with a trained palliative care clinician
* Questionnaires and an exit interview
* Chart Review

It is expected that about 70 participants currently receiving targeted therapy at Massachusetts General Hospital for lung cancer will take part in this research study: 10 patients in an open pilot study, followed by 60 patients in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* MGH Cancer Center patient
* Within 6 months of diagnosis of metastatic NSCLC with oncogenic driver mutation (EGFR, ALK, ROS1, RET)
* Receiving targeted therapy
* Ability to respond in English or Spanish

Exclusion Criteria:

* Cognitive impairment or serious mental illness that limits ability to provide informed consent
* Need for urgent palliative care or hospice referral
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of POISE - enrollment | 20 weeks
  ≥60% enrollment among eligible patientsamong patients in the POISE group
Feasibility of POISE - completion of all sessions among patients in intervention group | 20 weeks
  ≥70% completion of all sessions in the intervention arm
Feasibility of POISE - completion of surveys in both arms | 20 weeks
  ≥70% completion of all surveys in both arms

SECONDARY OUTCOMES:
Acceptability | 20 Weeks
  4-item measure of satisfaction and comfort with the intervention
Emotional coping with prognosis and prognostic awareness | 12 weeks
  Subscale of Prognostic Awareness Impact Scale
Emotional coping with prognosis and prognostic awareness | 20 weeks
  Subscale of Prognostic Awareness Impact Scale
Self efficacy | 12 weeks
  Self-Efficacy of Management of Chronic Disease 6-Item Scale asks patients to rate their confidence in managing symptoms and activities related to chronic disease on a 1-10 scale, ranging from 1 (not at all confident) to 10 (totally confident).
Self efficacy | 20 weeks
  Self-Efficacy of Management of Chronic Disease 6-Item Scale asks patients to rate their confidence in managing symptoms and activities related to chronic disease on a 1-10 scale
Documentation of Goals and Values | 20 weeks
  The investigators will apply a previously developed natural language processing/machine learning (ML) algorithm to palliative care and oncology notes from the study period in order to identify goals of care conversations using an inductive supervised ML classifier. Notes with a predicted probability of greater than 0.5 will be classified as containing goals of care documentation.

OTHER OUTCOMES:
Uncertainty tolerance | 12 weeks
  Intolerance of Uncertainty-Short Form is a 12-item questionnaire with descriptions about ability to tolerate uncertainty, using a Likert scale of agreement from 1 to 5, with lower scores indicating low intolerance of uncertainty and high scores indicating high intolerance of uncertainty.
Uncertainty tolerance | 20 weeks
  Intolerance of Uncertainty-Short Form is a 12-item questionnaire with descriptions about ability to tolerate uncertainty, using a Likert scale of agreement from 1 to 5, with lower scores indicating low intolerance of uncertainty and high scores indicating high intolerance of uncertainty.
Psychological Distress | 12 weeks
  Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire that contains two 7-item subscales assessing depression and anxiety symptoms during the past week, with higher scores indicating worse anxiety and depression.
Psychological Distress | 20 weeks
  Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire that contains two 7-item subscales assessing depression and anxiety symptoms during the past week, with higher scores indicating worse anxiety and depression.
Multidimensional quality of life | 12 weeks
  Functional Assessment of Cancer Therapy-Lung, a quality of life measure
Multidimensional quality of life | 20 weeks
  Functional Assessment of Cancer Therapy-Lung, a quality of life measure
Hope and goal setting | 12 weeks
  Adult Trait Hope Scale
Hope and goal setting | 20 weeks
  Adult Trait Hope Scale

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Petrillo, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Background] Richard HA, Sarathy R, Rabideau DJ, Feldman J, Cartagena L, Patel H, Sequist LV, Park E, Jackson V, Greer JA, Temel JS, Petrillo LA. Blended palliative and survivorship care intervention (POISE) for patients with metastatic oncogene-driven non-small cell lung cancer: study protocol for a pilot randomised controlled trial. BMJ Open. 2025 Aug 13;15(8):e098075. doi: 10.1136/bmjopen-2024-098075. PMID 40812801
- See also: Protocol paper — https://bmjopen.bmj.com/content/bmjopen/15/8/e098075.full.pdf